CLINICAL TRIAL: NCT02478060
Title: A Double-Blind, Randomised, Placebo-Controlled, Escalating, Multiple Dose Study in to Assess the Safety, Tolerability and Pharmacodynamic Effects of Birch-SPIRE
Brief Title: Birch-SPIRE Safety and Efficacy Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CB001
Record Dates: First submitted 2015-06-11; First posted 2015-06-23 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Rhinitis
Keywords: Allergy; Birch; Rhinitis; Rhinoconjuntivitis; SPIRE; Toleromune
MeSH Terms: conditions — Rhinitis; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): Birch-SPIRE or placebo, 2 weeks apart
  Interventions: Biological: Birch-SPIRE; Biological: Placebo
- Cohort 2 (Experimental): Birch-SPIRE or placebo, 2 weeks apart
  Interventions: Biological: Birch-SPIRE; Biological: Placebo
- Cohort 3 (Experimental): Birch-SPIRE or placebo, 2 weeks apart
  Interventions: Biological: Birch-SPIRE; Biological: Placebo
- Cohort 4 (Experimental): Birch-SPIRE or placebo, 2 weeks apart
  Interventions: Biological: Birch-SPIRE; Biological: Placebo
- Cohort 5 (Experimental): Birch-SPIRE or placebo, 2 weeks apart
  Interventions: Biological: Birch-SPIRE; Biological: Placebo

INTERVENTIONS:
Biological: Birch-SPIRE
Biological: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple administrations of Birch-SPIRE. To make a preliminary assessment on pharmacodynamic parameters and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 65 years;
* Minimum 1 year history of rhinitis with or without conjunctivitis on exposure to birch pollen
* Birch IgE ≥ 0.35 kU/L
* Positive skin prick test to whole birch allergen

Exclusion Criteria:

* Any past history of asthma
* FEV1 < 80% of predicted
* History of severe allergic reaction to birch allergen, severe drug allergy, severe angioedema or severe allergic reactions to food
* Acute phase skin response to whole birch allergen with a mean wheal diameter > 50mm
* Administration of adrenaline (epinephrine) is contraindicated
* History of severe drug allergy or anaphylactic reaction to food.
* History of any significant disease or disorder (e.g. immune system, pulmonary, cardiovascular, gastrointestinal, liver, renal, neurological, metabolic, malignant, psychiatric, major physical impairment, history of alcohol or drug abuse)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety of Birch-SPIRE administrations measured by Adverse Events | Up to 16 weeks after start of dosing

SECONDARY OUTCOMES:
Measurement of IgE as a Pharmacodynamic parameter | Up to 9 months after start of dosing
Conjunctival Provocation Test as a Pharmacodynamic parameter | Up to 9 months after start of dosing
Skin Prick Testing as a Pharmacodynamic parameter | Up to 9 months after start of dosing

OTHER OUTCOMES:
Allergy symptoms and allergy medication use during next Birch season | Up to 9 months after start of dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche Appliqué en Allergie de Québec, Québec, Quebec, Canada